CLINICAL TRIAL: NCT01409512
Title: Observational Study on the Effect of Anticholinergic on the Autonomic System in Women With OAB
Brief Title: Evaluation of Autonomic System Before and After Anticholinergic Treatment in Women With Overactive Bladder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dalia Kesner, Kupat Hulim Clalit
Other Study IDs: 117/2011
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Overactive Bladder
Keywords: Heart rate variability, anti cholinergic medication
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with OAB: Patients that will be diagnosed as having OAB syndrome by an urogynecologist based on their clinical symptoms (urinary urgency, with or without urinary urgency incontinence, urinary frequency or nocturia).
  Interventions: Procedure: ECG recording

INTERVENTIONS:
Procedure: ECG recording — At baseline and following 3 months on anticholinergic medications patients, ECG recording will be conducted.
  Other Names: Electro cardiogram recording

SUMMARY:
The aim of the study is to evaluate changes in autonomic nervous system following treatment with anticholinergic medication for OAB symptoms.

Heart variability as a measure of the functioning of the autonomic nervous system will be recorded before and three months following treatment with solifenacin succinate 10 mg daily.

DETAILED DESCRIPTION:
30 women with clinical diagnosis of overactive bladder will be recruited for the study. An ECG strip for fifteen minutes at rest will be recorded through a 12-bit analog/digital data acquisition card (National Instruments, Austin TX) with a sampling frequency of 200 Hz and stored in a computer for offline studies. The digitized ECG signals will than processed and analyzed via dedicated robust software to detect the R wave peaks. The R point of each QRS complex was defined and the interval between two consecutive R points (the R-R interval) was computed. All R-R intervals will be visually inspected and manually edited if necessary to exclude background noise and artifacts. The edited segments accounts for less than 1% in each patient. A "clean" 2-5-min segment (preferably unedited) will be used for the analyses. An autoregressive model with the order of 16 was will be used to estimate the power spectrum densities of HRV. The power spectra are quantified by measuring the area under the following frequency bands: low-frequency (LF) (0.04-0.15 Hz) known to represents sympathetic activity, and high-frequency (HF) (0.15-0.4 Hz) which represents parasympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of OAB

Exclusion Criteria:

1) stress urinary incontinence and voiding symptoms, 2) pregnancy, 3) pathological conditions that can interfere with the ANS, (e.g. coronary heart disease, heart failure, or other cardiac conditions, hypertension, neurological diseases or diabetes , 4) medications that can interfere with the ANS, including beta-receptor agonists or antagonists, antiarrhythmic agents or antihypertensive drugs, anticholinergic agents or adrenergic alpha-antagonists, tricyclic or serotoninergic antidepressants.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed as having OAB syndrome by an urogynecologist based on their clinical symptoms (urinary urgency, with or without urinary urgency incontinence, urinary frequency or nocturia).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Changes in heart variability following treatment with Solifenacin succinate 10 mg | 24 months

SECONDARY OUTCOMES:
Correlation between changes in clinical symptoms of OAB abd changes in heart rate variability | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowensrtein, MD, Study Chair — Rambam Health Care Campus
Locations (1):
- Zvolon Medical Center, Haifa, Israel

REFERENCES:
- [Background] Mehnert U, Knapp PA, Mueller N, Reitz A, Schurch B. Heart rate variability: an objective measure of autonomic activity and bladder sensations during urodynamics. Neurourol Urodyn. 2009;28(4):313-9. doi: 10.1002/nau.20641. PMID 19058189
- [Background] Liao WC, Jaw FS. A noninvasive evaluation of autonomic nervous system dysfunction in women with an overactive bladder. Int J Gynaecol Obstet. 2010 Jul;110(1):12-7. doi: 10.1016/j.ijgo.2010.03.007. Epub 2010 Apr 25. PMID 20423739
- [Background] Schiffers M, Sauermann P, Schurch B, Mehnert U. The effect of tolterodine 4 and 8 mg on the heart rate variability in healthy subjects. World J Urol. 2010 Oct;28(5):651-6. doi: 10.1007/s00345-010-0513-y. Epub 2010 Feb 7. PMID 20140437
- [Background] Hubeaux K, Deffieux X, Ismael SS, Raibaut P, Amarenco G. Autonomic nervous system activity during bladder filling assessed by heart rate variability analysis in women with idiopathic overactive bladder syndrome or stress urinary incontinence. J Urol. 2007 Dec;178(6):2483-7. doi: 10.1016/j.juro.2007.08.036. Epub 2007 Oct 15. PMID 17937953